CLINICAL TRIAL: NCT00000919
Title: Study of Protease Inhibitor and/or Non-Nucleoside Reverse Transcriptase Inhibitor With Dual Nucleosides in Initial Therapy of HIV Infection
Brief Title: A Study to Evaluate Various Combinations of Anti-HIV Medications to Treat Early HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 384; 11343 (Registry Identifier: DAIDS ES); AACTG A5005s; AACTG A5006s; AACTG A5007s; AACTG A5031s; AACTG 731
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; lamivudine, zidovudine drug combination; Ritonavir; Hydroxyurea; abacavir; amprenavir; Nelfinavir; efavirenz; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine/Zidovudine
Drug: Ritonavir
Drug: Hydroxyurea
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare the effectiveness of various combinations of anti-HIV drugs in HIV-positive men and women. Patients receive specific combinations of 3 or 4 of the following 6 drugs: didanosine (ddI), stavudine (d4T) efavirenz (EFV), nelfinavir (NFV), lamivudine (3TC), or zidovudine (ZDV).

Anti-HIV therapy is effective in preventing the spread of HIV in the body. However, patients often experience unpleasant side effects and have difficulties following the dosing schedule. This study looks for combinations of anti-HIV drugs ("cocktails") which will be the most effective with the fewest problems.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy, though effective in the suppression of HIV proliferation, is often complicated by difficulties with adherence and drug toxicity. Various combinations of highly active antiretroviral therapy exist; all have proved efficacious in related trials. The question addressed in this trial is which combination of antiretroviral "cocktails" provides the single greatest advantage in preventing the spread of HIV in the body. In effect, which therapy provides the greatest benefit with the fewest complications.

Step 1: Patients are randomized to 1 of 6 arms:

Arm A: didanosine (ddI), stavudine (d4T), efavirenz (EFV), and nelfinavir (NFV) placebo.

Arm B: ddI, d4T, EFV placebo, and NFV. Arm C: lamivudine (3TC)/zidovudine (ZDV), EFV, and NFV placebo. Arm D: 3TC/ZDV, EFV placebo, and NFV. Arm E: ddI, d4T, EFV, and NFV. Arm F: 3TC/ZDV, EFV, and NFV. Patients with virologic failure on 2 successive measurements or study-drug intolerance discontinue their randomized study therapy and proceed to Step 2. [AS PER AMENDMENT 7/5/00: Patients must switch regimens as soon as possible after confirmation of virologic failure to prevent development of drug resistance.]

Step 2:

Arm A: Patients receive treatment as in Arm D of Step 1. Arm B: Patients receive treatment as in Arm C of Step 1. Arm C: Patients receive treatment as in Arm B of Step 1. Arm D: Patients receive treatment as in Arm A of Step 1. Arms A, B, C, and D: Patients who fail Step 2 treatment proceed to Step 3. Arms E and F: Patients with virologic failure on Step 1 proceed immediately to Step 3.

Step 3 (salvage therapy):

Arm A, B, C, and D: Patients receive indinavir (IDV), amprenavir (APV), ddI, and hydroxyurea (HU).

[AS PER AMENDMENT 7/5/00: Patients now receive treatment on Regimen 1, 2, 3, 4, 5, or 6. Regimen 1 consists of IDV, ritonavir (RTV), ddI, and HU. Regimen 2 consists of APV, RTV, ddI, and HU. Regimen 3 consists of IDV, RTV, abacavir (ABC), and 3TC/ZDV. Regimen 4 consists of APV, RTV, ABC, and 3TC/ZDV. Regimen 5 consists of IDV, RTV, ABC, d4T, and 3TC. Regimen 6 consists of APV, RTV, ABC, d4T, and 3TC.] Arm E: Patients receive IDV, APV, and 3TC/ZDV. [AS PER AMENDMENT 7/5/00: Patients now receive treatment on Regimen 7 or 8. Regimen 7 consists of IDV, RTV, and 3TC/ZDV. Regimen 8 consists of APV, RTV, and 3TC/ZDV.] Arm F: Patients receive IDV, APV, ddI, and d4T. [AS PER AMENDMENT 7/5/00: Patients now receive treatment on Regimen 9 or 10. Regimen 9 consists of IDV, RTV, ddI, and d4T. Regimen 10 consists of APV, RTV, ddI, and d4T.] [AS PER AMENDMENT 7/5/00: Patients already enrolled in Step 3 before site registration to Version 4.0 of this protocol have the option of receiving 1 of the appropriate new Step 3 regimens as outlined above or staying on their originally assigned Step 3 therapy.] [AS PER AMENDMENT 3/21/01: If virologic failure on Step 1 or 2 is confirmed, then HIV-1 RNA genotype resistance testing (in real-time, if possible) is performed. Patients receive 1 of the Step 3 drug regimens based on the results of the resistance testing.] Patients may co-enroll in metabolic, pharmacologic, immunologic, or adherence substudies.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

[Required: AS PER AMENDMENT 7/5/00:

* Chemoprophylaxis for Pneumocystis carinii pneumonia if CD4+ cell count is less than or equal to 200 cells/mm3.]

[Suggested as an alternative agent for chemoprophylaxis against Mycobacterium avium complex:

* Azithromycin.]

[Allowed: AS PER AMENDMENT 7/5/00:

* Topical and oral antifungal agents. Oral itraconazole may be administered concurrently with IDV if the dose of IDV is reduced to 600 mg every 8 hours.
* Treatment, maintenance, or chemoprophylaxis for opportunistic infections, as clinically indicated unless otherwise prohibited by the protocol.
* All antibiotics, as clinically indicated unless otherwise prohibited by the protocol.
* Systemic corticosteroid use for 21 days or less for acute problems, as medically indicated.
* Recombinant erythropoietin (rEPO, epoetin alfa, Epogen, epoetin beta, Marogen), granulocyte colony-stimulating factor (G-CSF, filgrastim, Neupogen), and granulocyte-macrophage colony-stimulating factor (GM-CSF, Regramostim).
* Regularly prescribed medications, such as antipyretics, analgesics, allergy medications, antidepressants, sleep medications, oral contraceptives, megestrol acetate (Megace), testosterone, or any other medications, as medically indicated unless otherwise prohibited by the protocol. NOTE: Due to the possibility that study medications may alter the effectiveness of oral contraceptives or depoprogesterone, these agents must not be used as the sole form of birth control, because the role of some study medications on the effectiveness of these methods has not yet been established.
* Alternative therapies, such as vitamins.
* Medications requiring low gastric pH if not administered at the same time as buffered ddI. Patients taking these agents should do so at least 2 hours before ddI.]
* Vaccinations, if administered at least 2 weeks prior to an HIV RNA viral load evaluation.

[Allowed with caution: AS PER AMENDMENT 7/5/00:

* Oral ketoconazole with IDV.

Medications that interact with PIs as substrates, inhibitors, or inducers, including, but not limited to:

* allopurinol, alprazolam, amitriptyline, atorvastatin, bupropion, carbamazepine, cerivastatin, chlorpheniramine, chlorpromazine, chlorzoxazone, cimetidine, clarithromycin, clofibrate, clorazepate, clozapine, codeine, dapsone, desipramine, diazepam, diltiazem, disopyramide, encainide, erythromycin, estazolam, estrogens and progesterones, fluoxetine, flurazepam, fluvastatin, glucocorticoids, hypericum perforatum (St. John's wort), imipramine, isoniazid, itraconazole, ketoconazole, labetalol, lamotrigine, lidocaine, lovastatin, mexiletine, morphine, naloxone, nefazodone, nifedipine, nortriptyline, opioids, oxazepam, pentazocine, phenobarbital, phenytoin, promethazine, propofol, propranolol and other beta blockers, sildenafil, simvastatin, temazepam, T3 (thyroid hormone), warfarin, valproic acid, and zolpidem.
* Drugs with high protein-binding properties, nephrotoxic drugs, and opiate agonists (e.g., methadone or buprenorphine).]

NOTE:

* Refer to package insert for potential drug interactions with IDV, RTV, NFV, or APV that may require therapeutic drug monitoring and/or adjustment of concomitant medications.]

[Allowed with extreme caution:

* AS PER AMENDMENT 7/5/00:

ddI, as clinically indicated in patients with known risk factors, including, but not limited to, alcohol abuse, morbid obesity, hypertriglyceridemia, cholelithiasis, endoscopic retrograde cholangiopancreatography, use of medications known to cause pancreatitis (e.g., pentamidine) and use of medications known or thought to increase exposure to ddI (e.g., HU, allopurinol).]

Concurrent Treatment:

[Allowed:

* AS PER AMENDMENT 7/5/00:

Acupuncture and visualization techniques.]

Patients must have:

* HIV infection, as documented by any licensed ELISA test kit and confirmed by either Western blot, HIV culture, HIV antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA at any time prior to study entry.
* Plasma HIV-1 RNA of 500 copies/ml or more, confirmed by the Roche Amplicor assay only and performed within 60 days [AS PER AMENDMENT 5/5/99:
* 70 days] of study entry by any certified laboratory.
* Inclusion laboratory parameters, documented within 14 days prior to study entry (see lab values).

[AS PER AMENDMENT 9/9/99:

* Co-enrollment on ACTG A5005s (Metabolism Substudy) is required for patients enrolling under Version 3.0 of ACTG 384.]

Risk Behavior:

[Allowed with caution:

* AS PER AMENDMENT 7/5/00:

Alcoholic beverages.]

Exclusion Criteria

Co-existing Condition:

Patients with the following condition are excluded:

AIDS-related malignancy other than minimal Kaposi's sarcoma.

Concurrent Medication:

[Excluded:

* AS PER AMENDMENT 7/5/00:
* Chronic systemic corticosteroids.
* For Steps 1 and 2, all antiretroviral therapies other than study medications. For step 3, contact the team to discuss potential addition or substitution with off-study antiretroviral medications.
* Investigational drugs without specific approval from the study chairs.
* Neurotoxic and pancreatotoxic drugs.
* Systemic cytotoxic chemotherapy.
* Amiodarone, astemizole, bepridil, cisapride, cholestyramine, ergot and ergot derivatives, flecainide, ganciclovir, interferon alfa, midazolam (unless used for sedation on ACTG 723), pimozide, propafenone, propoxyphene, quinidine, ribavirin, rifampin, sucralfate, terfenadine, and triazolam.
* Rifabutin for patients on RTV in Step 3 and for patients on Steps 1 and 2 because of the contradictory effects of EFV and NFV on plasma rifabutin levels. If a patient on Step 1 or 2 requires treatment with rifabutin after coming on the study, the team must be notified.
* Alpha tocopherol (vitamin E) supplementation since vitamin E is contained in the soft gelatin capsule formulation of APV.
* ddI concurrently with IV pentamidine.
* Herbal medications.]

Patients with the following prior conditions are excluded:

* Pancreatitis within 3 years of study entry.
* Current peripheral neuropathy grade 2 or greater or history of peripheral neuropathy grade 3 or greater.
* Documented or suspected acute hepatitis within 30 days prior to study entry.
* Unexplained temperature above 38.5 C for any 7 days or chronic diarrhea (defined as more than 3 liquid stools per day persisting for more than 15 days) within 30 days prior to study entry.
* Any previous hypersensitivity to study drugs or their components.

Prior Medication:

Excluded:

* Receipt within 30 days of erythropoietin, G-CSF, or GM-CSF.
* Treatment within 14 days of study entry with any of the following:
* amiodarone, astemizole, cisapride, ergot or ergot derivatives, ketoconazole, midazolam, propoxyphene, quinidine, rifampin, terfenidine, or triazolam.
* Prior antiretroviral therapy for 7 days or more, including protease inhibitors (PIs), nucleoside reverse transcriptase inhibitors (NRTIs), and nonnucleoside reverse transcriptase inhibitors (NNRTIs). [AS PER AMENDMENT 5/5/99:
* Systemic ketoconazole or itraconazole, intravenous pentamidine, and rifabutin are prohibited. Midazolam is allowed for sedation in patients participating on ACTG 723.]
* Any vaccination within 14 days prior to study entry.
* Any immunomodulator or investigational therapy within 30 days prior to study entry.

[AS PER AMENDMENT 5/5/99:

* 6. Rifabutin is discouraged.]

Prior Treatment:

Excluded:

* Acute therapy for an infection or other medical illness within 14 days prior to study entry.

[AS PER AMENDMENT 5/5/99:

* Acute therapy for a serious infection or other serious medical illness that is potentially life-threatening and requires systemic therapy and/or hospitalization within 14 days of study entry. Patients with Pneumocystis carinii pneumonia must have completed acute therapy at least 7 days prior to entry and be clinically stable. Patients with other serious infection or serious medical illness who must continue chronic therapy must have completed at least 14 days of therapy prior to entry and be clinically stable. Patients with all other infections or medical illnesses must have completed therapy, or at least 14 days of maintenance therapy, prior to entry and be clinically stable (restrictions do not apply to oral and vaginal candidiasis, mucocutaneous herpes simplex infection, and minor skin conditions).]

Risk Behavior:

Excluded:

* Possible current substance abuse that could prevent compliance with the study medication.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shafer, Study Chair; Gregory Robbins, Study Chair
Locations (80):
- United States (63):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - Marin County Specialty Clinic, San Rafael, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Hosp, Washington D.C., District of Columbia
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Emory Hemo Comp Evaluation Clinic / East TN Comp Hemo Ctr, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Med Ctr Hosp, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Manhattan Veterans Administration / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med Ctr, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington
- Italy (14):
  - Azienda Ospedaliera Umberto I, Ancona
  - Ospedale S Orsola, Bologna
  - Spedali Civili - Carosi, Brescia
  - Spedali Civili Cadeo, Brescia
  - Archispedale S Anna, Ferrara
  - Universita di Genova, Genova
  - Ospedale Luigi Cacco Moroni, Milan
  - Ospedale Luigi Sacco Cargnel, Milan
  - Azienda Ospedaliera di Parma, Parma
  - IRCCS Policlinico S Matteo Filice, Pavia
  - IRCCS Policlinico S Matteo Minoli, Pavia
  - Archispedale S Maria Nuova, Reggio Emilia
  - Universita di Roma - Delia, Roma
  - Ospedale Civile Maggiore, Verona
- Univ of Puerto Rico, San Juan, Puerto Rico
- Country not given (2):
  - Azienda USL di Piacenza
  - Francesco Leoncini

REFERENCES:
- [Background] Smeaton LM, DeGruttola V, Robbins GK, Shafer RW. ACTG (AIDS Clinical Trials Group) 384: a strategy trial comparing consecutive treatments for HIV-1. Control Clin Trials. 2001 Apr;22(2):142-59. doi: 10.1016/s0197-2456(00)00126-4. PMID 11306153
- [Background] Dube MP, Zackin R, Tebas P, et al. Prospective study of regional body composition in antiretroviral-naive subjects randomized to receive zidovudine+lamivudine or didanosine+stavudine combined with nelfinavir, efavirenz, or both: A5005s, a substudy of ACTG 384. Antiviral Ther. 2002;7:L18. Abstract 27.
- [Background] Smith PF, Robbins G, Shafer R, Wu H, Yu S, Hirsch M, Merigan T, Morse GD, ACTG 384 Study Team. Effect of Efavirenz on the Pharmacokinetics of Nelfinavir and M8 in Naïve, HIV-infected Patients Receiving Long-term HAART Therapy. 10th Conference on Retroviruses and Oppurtunistic Infections. Feb 2003. Abstract 148.
- [Result] Shafer RW, Smeaton LM, Robbins GK, De Gruttola V, Snyder SW, D'Aquila RT, Johnson VA, Morse GD, Nokta MA, Martinez AI, Gripshover BM, Kaul P, Haubrich R, Swingle M, McCarty SD, Vella S, Hirsch MS, Merigan TC; AIDS Clinical Trials Group 384 Team. Comparison of four-drug regimens and pairs of sequential three-drug regimens as initial therapy for HIV-1 infection. N Engl J Med. 2003 Dec 11;349(24):2304-15. doi: 10.1056/NEJMoa030265. PMID 14668456
- [Result] Robbins GK, De Gruttola V, Shafer RW, Smeaton LM, Snyder SW, Pettinelli C, Dube MP, Fischl MA, Pollard RB, Delapenha R, Gedeon L, van der Horst C, Murphy RL, Becker MI, D'Aquila RT, Vella S, Merigan TC, Hirsch MS; AIDS Clinical Trials Group 384 Team. Comparison of sequential three-drug regimens as initial therapy for HIV-1 infection. N Engl J Med. 2003 Dec 11;349(24):2293-303. doi: 10.1056/NEJMoa030264. PMID 14668455
- [Result] Reynolds NR, Testa MA, Marc LG, Chesney MA, Neidig JL, Smith SR, Vella S, Robbins GK; Protocol Teams of ACTG 384, ACTG 731 and A5031s. Factors influencing medication adherence beliefs and self-efficacy in persons naive to antiretroviral therapy: a multicenter, cross-sectional study. AIDS Behav. 2004 Jun;8(2):141-50. doi: 10.1023/B:AIBE.0000030245.52406.bb. PMID 15187476
- [Result] Hulgan T, Haas DW, Haines JL, Ritchie MD, Robbins GK, Shafer RW, Clifford DB, Kallianpur AR, Summar M, Canter JA. Mitochondrial haplogroups and peripheral neuropathy during antiretroviral therapy: an adult AIDS clinical trials group study. AIDS. 2005 Sep 2;19(13):1341-9. doi: 10.1097/01.aids.0000180786.02930.a1. PMID 16103764
- [Result] Smith PF, Robbins GK, Shafer RW, Wu H, Yu S, Hirsch MS, Merigan TC, Park JG, Forrest A, Fischl MA, Morse GD; ACTG 384-5006 Team. Pharmacokinetics of nelfinavir and efavirenz in antiretroviral-naive, human immunodeficiency virus-infected subjects when administered alone or in combination with nucleoside analog reverse transcriptase inhibitors. Antimicrob Agents Chemother. 2005 Aug;49(8):3558-61. doi: 10.1128/AAC.49.8.3558-3561.2005. PMID 16048984
- [Result] Haas DW, Smeaton LM, Shafer RW, Robbins GK, Morse GD, Labbe L, Wilkinson GR, Clifford DB, D'Aquila RT, De Gruttola V, Pollard RB, Merigan TC, Hirsch MS, George AL Jr, Donahue JP, Kim RB. Pharmacogenetics of long-term responses to antiretroviral regimens containing Efavirenz and/or Nelfinavir: an Adult Aids Clinical Trials Group Study. J Infect Dis. 2005 Dec 1;192(11):1931-42. doi: 10.1086/497610. Epub 2005 Nov 1. PMID 16267764
- [Result] Gandhi RT, Spritzler J, Chan E, Asmuth DM, Rodriguez B, Merigan TC, Hirsch MS, Shafer RW, Robbins GK, Pollard RB; ACTG 384 Team. Effect of baseline- and treatment-related factors on immunologic recovery after initiation of antiretroviral therapy in HIV-1-positive subjects: results from ACTG 384. J Acquir Immune Defic Syndr. 2006 Aug 1;42(4):426-34. doi: 10.1097/01.qai.0000226789.51992.3f. PMID 16810109
- [Result] Marc LG, Testa MA, Walker AM, Robbins GK, Shafer RW, Anderson NB, Berkman LF; ACTG Data Analysis Concept Sheet Study Team. Educational attainment and response to HAART during initial therapy for HIV-1 infection. J Psychosom Res. 2007 Aug;63(2):207-16. doi: 10.1016/j.jpsychores.2007.04.009. PMID 17662759
- [Derived] Li B, Veturi Y, Verma A, Bradford Y, Daar ES, Gulick RM, Riddler SA, Robbins GK, Lennox JL, Haas DW, Ritchie MD. Tissue specificity-aware TWAS (TSA-TWAS) framework identifies novel associations with metabolic, immunologic, and virologic traits in HIV-positive adults. PLoS Genet. 2021 Apr 26;17(4):e1009464. doi: 10.1371/journal.pgen.1009464. eCollection 2021 Apr. PMID 33901188
- [Derived] Lok JJ, Hunt PW, Collier AC, Benson CA, Witt MD, Luque AE, Deeks SG, Bosch RJ. The impact of age on the prognostic capacity of CD8+ T-cell activation during suppressive antiretroviral therapy. AIDS. 2013 Aug 24;27(13):2101-10. doi: 10.1097/QAD.0b013e32836191b1. PMID 24326304
- [Derived] Lok JJ, Bosch RJ, Benson CA, Collier AC, Robbins GK, Shafer RW, Hughes MD; ALLRT team. Long-term increase in CD4+ T-cell counts during combination antiretroviral therapy for HIV-1 infection. AIDS. 2010 Jul 31;24(12):1867-76. doi: 10.1097/QAD.0b013e32833adbcf. PMID 20467286